CLINICAL TRIAL: NCT02037867
Title: The Stratification of Liver Disease in the Community Using Fibrosis Biomarkers
Brief Title: Nottingham Community Liver Biomarkers Cohort
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 13029; 13/EM/0123 (Other: Research Ethics Committee (East Midlands - Leicester))
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Chronic Liver Disease; Alcohol Use Disorder; Type 2 Diabetes; Persistently Elevated ALT; Obesity
Keywords: alcohol; type 2 diabetes; ALT; abnormal liver enzymes; hepatic fibrosis; cirrhosis
MeSH Terms: conditions — Alcoholism; Diabetes Mellitus, Type 2; Obesity; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Serum, whole blood and urine samples stored a -80 degrees Celsius.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients identified with one of the below chronic liver disease risk factors and undergoing community liver disease stratification using fibrosis biomarkers:
  * Hazardous alcohol use (>14 units per week in females, >21 units per week in males, alcohol AUDIT score >=8 or read code relevant to alcohol abuse on GP system)
  * Type 2 Diabetes
  * Obesity
  * Persistently raised serum ALT level, negative liver serology, and absence of above 2 risk factors
  Interventions: Device: Fibrosis Biomarkers

INTERVENTIONS:
Device: Fibrosis Biomarkers — Liver disease stratification with liver stiffness scan (Transient Elastography) Analysis of diagnostic performance of serum fibrosis markers (as listed above) Whole blood samples obtained for DNA analysis
  Other Names: AST:ALT ratio, APRI, BARD score, ELF Score, FIB4, NAFLD Fibrosis Score,Transient Elastography

SUMMARY:
Deaths due to advanced liver scarring (liver cirrhosis) continue to increase, and liver disease is now the 3rd leading cause of premature death in the United Kingdom. The majority of liver disease is lifestyle related (alcohol, obesity and associated type 2 diabetes, injecting drug use) and therefore reversible if caught at a precirrhosis stage. However, current liver function blood tests are poor inadequate, and subsequently a large burden of liver disease is currently missed.

A variety of noninvasive liver biomarkers (blood and imaging tests) have been developed which identify liver disease accurately at earlier stages of scarring. The identification of liver disease in the community, where previous studies have discovered a large burden of previously unidentified but significant liver disease, is therefore a feasible place to develop new liver disease investigation pathways using these noninvasive markers.

In collaboration with the Department of Health, Nottingham University Hospitals have commenced a pilot community liver disease pathway in two General Practices in Nottingham in February 2012. Patients with liver risk factors (hazardous alcohol use, obesity or type 2 diabetes)are invited to take part in the pathway. Patients undergo a simple blood test (AST:ALT ratio and BARD score), with a high test result requiring referral for a liver stiffness scan (Fibroscan)which is performed in the community setting. High threshold scan values are reviewed by a consultant liver specialist in a community liver clinic. Preliminary findings show that the pathway accurately identifies patients with early liver scarring and previously unidentified significant liver disease. The participating General Practitioners have also noted a striking number of patients finally engaging in important lifestyle changes following pathway implementation. A second phase of the pilot pathway, in 2 Inner City General Practices with a total practice population of c.14,000 patients commenced in June 2013.

We have subsequently designed this cohort study, where pilot participants will be consented for follow up over a long period. We will assess future liver-related and cardiovascular events (including death), and perform qualitative patient interviews to assess the reasons for and persistence of lifestyle changes after liver disease investigation. We hypothesize that stratification of liver disease in the community will unearth a significant amount of previously undetected but significant chronic liver disease. Moreover, we will evaluate whether stratification of liver disease using these tests predicts future liver and cardiovascular disease and death, and whether stratification has an impact on patient's future lifestyle choices.

DETAILED DESCRIPTION:
Objectives:

1. To establish a community based cohort with risk factors for liver disease and stratification for liver disease severity using non-invasive biomarkers.
2. To establish the incidence of liver and cardiovascular morbidity and mortality in a community cohort.
3. To explore the quantitative and qualitative indicators to potential alterations in patient lifestyle following stratification of liver disease to inform future intervention development.
4. To evaluate novel blood markers of liver fibrosis and cirrhosis on a large cohort of primary care patients

Study Configuration:

Longitudinal Cohort Study with long-term follow up

Setting:

Primary Care, Nottingham

Number of Participants:

Prospective and consecutive recruitment in the East Midlands - approximately 500 patients per annum over a 4 year cohort inception period. Total anticipated cohort size 2,000 participants.

Description of Interventions:

* Serum blood sampling (AST:ALT ratio, and serum stored for future liver biomarker development)
* Transient Elastography (Fibroscan)
* Qualitative Interviews (limited to approximately 30 patients)
* Consent to longitudinal data follow-up and approach for future lifestyle intervention trials - consenting patients will be tagged on MRIS database.

Duration of Study:

48 month cohort inception with long term longitudinal follow up of cardiovascular and liver related outcomes and mortality data.

Outcome Measures:

1. Incidence of liver (cirrhosis) and cardiovascular disease (symptomatic coronary or cerebrovascular disease).
2. All cause morbidity and mortality.
3. Quantitative and qualitative lifestyle measures (including body mass index, exercise levels, alcohol consumption).

Patients who decide to participate in the community cohort will not be required to perform any specific actions or attend study visits (unless for the reasons stated below). Usual clinical care (both liver-related and non-liver related) will continue during the study period.

Patients will consent to long term longitudinal data follow-up using the Medical Research Information Service (MRIS) database. All patients enrolled in the community cohort will be prospectively tagged on MRIS. In particular, the investigators will request individual patient alerts on MRIS concerning prevalent cardiovascular disease events (angina, myocardial infarction and stroke), liver cirrhosis and cause of death.

Patients will consent to undertake qualitative research to evaluate the process of community stratification. A purposeful sample of patients completing the community biomarkers pathway will be invited to participate in qualitative follow up of their experiences of the pathway and any subsequent lifestyle change. A researcher, trained in qualitative research methods, will perform a semi-structured interview, which will assess any lifestyle changes occurring following liver pathway stratification. Specifically, changes in alcohol consumption, diet and exercise will be explored and evaluated, with assessment of the relationship to liver pathway stratification (both investigation results and lifestyle advice offered during the pathway). Interviews will performed either face-to-face, in which case this will be performed at the Nottingham Digestive Diseases Biomedical Research Unit, or over the telephone - in all cases voice recording will occur to allow analysis of information provided. An example interview proforma to be utilized for these qualitative interviews has been provided separately.

Patients will be consented to donate biosamples (including blood and urine) to the Nottingham Health Sciences Biobank on inception into the cohort. An appointment will be made at the NIHR Nottingham Digestive Diseases Biomedical Research Unit for witnessed written consent and to allow donation of biosamples. Samples will be collected by trained research nurses, who also form part of the research team. These biosamples will be utilized for future research into novel biomarkers of liver and cardiovascular disease, including proteomics and metabonomics. Where participants do not agree to the future use of the samples they will be destroyed in accordance with the Human Tissue Act, 2004.

In the future, the investigators will plan trials assessing novel exercise and dietary interventions, and subsequent effects on patient lifestyle parameters and future cardiovascular risk. Patients forming the community cohort will consent for contact regarding these future trials; however individual trials will be subject to their own ethical approval and written consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or over (male or female) with primary risk factor for liver disease:

  * Hazardous alcohol use (>14 units/week for women, >21 units/week for men)
  * Type 2 Diabetes
  * Obesity
  * Persistently elevated ALT with normal liver serology

Exclusion Criteria:

* Active malignancy at study enrolment
* Inability to provide informed consent for study enrolment
* Known presence of histologically proven liver disease prior to pilot pathway participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A Primary Care database search (Systmone, TPP)will be performed to identify patients eligible for study (see inclusion criteria) in the discrete patient populations.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-05; Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Liver and cardiovascular-related mortality | 20 years
  Death recorded as resulting from cardiovascular or liver-related causes

SECONDARY OUTCOMES:
Liver Cirrhosis | 20 years
  Incidence of compensated and decompensated cirrhosis diagnosis during the study period.
Cardiovascular Disease | 20 years
  Incidence of cardiovascular disease events(defined as symptomatic coronary or cerebrovascular disease)during the study period.
All-cause mortality | 20 years
  Recording of any death during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Neil Guha, MRCP, PhD, Principal Investigator — University of Nottingham
Locations (1):
- NIHR Nottingham Digestive Diseases Biomedical Research Unit, Nottingham, Notts, United Kingdom

REFERENCES:
- [Derived] Bradley CR, Cox EF, Palaniyappan N, Aithal GP, Francis ST, Guha IN. Variability of noninvasive MRI and biological markers in compensated cirrhosis: insights for assessing disease progression. Eur Radiol Exp. 2022 Oct 24;6(1):52. doi: 10.1186/s41747-022-00303-y. PMID 36274113
- [Derived] Tanajewski L, Harris R, Harman DJ, Aithal GP, Card TR, Gkountouras G, Berdunov V, Guha IN, Elliott RA. Economic evaluation of a community-based diagnostic pathway to stratify adults for non-alcoholic fatty liver disease: a Markov model informed by a feasibility study. BMJ Open. 2017 Jul 5;7(6):e015659. doi: 10.1136/bmjopen-2016-015659. PMID 28679676
- [Derived] Harman DJ, Ryder SD, James MW, Jelpke M, Ottey DS, Wilkes EA, Card TR, Aithal GP, Guha IN. Direct targeting of risk factors significantly increases the detection of liver cirrhosis in primary care: a cross-sectional diagnostic study utilising transient elastography. BMJ Open. 2015 May 3;5(4):e007516. doi: 10.1136/bmjopen-2014-007516. PMID 25941185
- See also: Nottingham Digestive Disease Biomedical Research Unit — http://www.nddcbru.org.uk/